CLINICAL TRIAL: NCT03982225
Title: A Multicenter, Randomized, Subject-assessor Blind, Placebo Controlled Phase Ⅱ Study to Determine the Optimal Dose of AYP-101 S.C. Injection for the Reduction of Submental Fat
Brief Title: Evaluate the Efficacy and Safety of Polyene Phosphatidylcholine Injection (AYP-101) for the Reduction of Submental Fat
Acronym: AYP-101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AMIpharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AYP-101-201
Record Dates: First submitted 2019-06-05; First posted 2019-06-11 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Moderate or Severe Submental Fullness
Keywords: Apoptosis; Lipolysis; Fat reduction; Submental fat; Polyene Phosphatidylcholine
MeSH Terms: conditions — Lymphoma, Follicular | interventions — polyene phosphatidylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2.5% Polyene Phosphatidylcholine Injection 0.2 mL/1.0 cm (Experimental): Participants receive 2.5% polyene phosphatidylcholine administered in 0.2 mL injections, 1.0 cm apart, up to 10.0 ml per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Polyene phosphatidylcholine injection
- 5.0% Polyene Phosphatidylcholine Injection 0.2 mL/1.0 cm (Experimental): Participants receive 5.0% polyene phosphatidylcholine administered in 0.2 mL injections, 1.0 cm apart, up to 10.0 ml per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Polyene phosphatidylcholine injection
- 5.0% Polyene Phosphatidylcholine Injection 0.4 mL/1.0 cm (Experimental): Participants receive 5.0% polyene phosphatidylcholine administered in 0.4 mL injections, 1.0 cm apart, up to 20.0 ml per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Polyene phosphatidylcholine injection
- Placebo 0.2 mL/1.0 cm (Placebo Comparator): Participants receive placebo administered in 0.2 mL injections, 1.0 cm apart, up to 10.0 ml per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyene phosphatidylcholine injection — Formulated as an injectable solution containing Polyene Phosphatidylcholine at two concentration of 25 mg/mL and 50 mg/mL.
  Other Names: AYP-101
  Arms: 2.5% Polyene Phosphatidylcholine Injection 0.2 mL/1.0 cm; 5.0% Polyene Phosphatidylcholine Injection 0.2 mL/1.0 cm; 5.0% Polyene Phosphatidylcholine Injection 0.4 mL/1.0 cm
Drug: Placebo — Phosphate buffered saline placebo for injection
  Arms: Placebo 0.2 mL/1.0 cm

SUMMARY:
Phase 2 trial to evaluate the safety and potential efficacy of three concentration of polyene phosphatidylcholine injection (AYP-101) compared to placebo for the reduction of submental fat.

DETAILED DESCRIPTION:
This study is to determine the optimal dose and evaluate safety and efficacy of Polyene Phosphatidylcholine S.C injection (AYP-101) for the reduction of Submental Fat (SMF) who wish improvement in the appearance of moderate to severe convexity or fullness associated with SMF in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female over 19 and under 65 years old.
2. Submental fat graded by the investigator as 2 or 3 using the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and graded by the subject as 2 or 3 using the Patient-Reported Submental Fat Rating Scale (PR-SMFRS) as determined on Visit 1.
3. Dissatisfaction with the submental area expressed by the subject as a rating of 0, 1, or 2 using the Subject Self Rating Scale (SSRS) as determined on Visit 1.
4. Stable weight over the last 6 months (body weight change within +/- 5kg), subject who should refrain from exercise and diet that may affect the study results, and who agreed to remain it for the study period.
5. Signed informed consent obtained before any study-specific procedure is performed.

Exclusion Criteria:

1. Allergic to beans or medical devices which used in this clinical trial (sterile oil pan, alcohol swab, grid pad, needle, etc.).
2. Hypersensitivity to the components of the clinical drug, lidocaine or acetaminophen.
3. Central, endocrine, or hereditary obesity (BMI 35kg/m2 or more).
4. Unable to undergo MRI by neurosis or general weakness.
5. History of any treatment (orthognathic surgery, suction lipectomy, Polyene Phosphatidylcholine (PPC) injection) in the neck or chin area.
6. History of any treatment such as massotherapy, carboxy, laser surgery, acupuncture needle, filler, chemical peeling, a botox surgery within 1 year before screening.
7. Inflammation, scars or surgery on the injection area.
8. Judged to be unsuitable subject for the clinical trials; ① Abnormal or sagging skin, ② Noticeable platysma band under the chin area, ③ Less or short chin than normal.
9. Chin or neck disease that are considered to have an impact on the clinical trial such as lymphadenopathy.
10. History of or present symptoms of dysphagia.
11. Heart disease (cardiac insufficiency, angina, cardiac infarction) or stroke within 6 months before screening.
12. Requiring treatment of joint inflammation or a lung disease.
13. Uncontrolled hypertension (systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 110 mmHg) or type 2 diabetes mellitus (HbA1c> 9%).
14. Type 1 diabetes mellitus who needs insulin treatment.
15. Autoimmune disorder as well as those who takes immunodepressant drugs.
16. Hemostatic disorder or those who takes anticoagulant drug such as warfarin and clopidogrel.
17. Thyromegaly, thyrotoxicosis, or HIV-positive.
18. Diagnosed with malignant tumor within the last 5 years.
19. Severe renal dysfunction (serum creatinine > 2.0 mg/dl) or severe dyshepatia (ALT, aspartate aminotransferase(AST), alkaline phosphatase > maximum rate of normality x 2.5).
20. History of serious psychiatric disease (Depression, schizophrenia, epilepsy, alcoholism, drug addiction, anorexia, anorexia nervosa, etc.).
21. History of taken a drug that can affect body weight or lipid metabolism such as anorectic agent, steroids, thyroid hormones, amphetamine, cyproheptadine, phenothiazine, or drugs that affect absorption, metabolism, and excretion within 3 months before screening.
22. History of other clinical trial studies within 3 months before screening.
23. Women who are pregnant, breastfeeding, having pregnancy plan, or did not agreed to the contraception (contraceptive pills, contraceptive hormones, intrauterine contraceptive device, spermicide, condoms etc.).
24. Judged to be unsuitable subject for the clinical trials.
25. No or unable to using Smart phone to fill in the e-Pro.
26. Artificial or cavity teeth filled with metallic material (iron, gold, amalgam, cobalt, titanium) which makes misinterpret MRI.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved a Composite 1-grade Response with Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) Compared to the Baseline | Baseline and 12 weeks after last treatment
  A composite 1-grade response is defined as at least a 1-grade improvement from Baseline on both the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) is evaluated by independent assessor and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) using the following scale:
  0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved a Composite 1-grade Response with Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) Compared to the Baseline | Baseline and 12 weeks after last treatment
  The CR-SMFRS is defined as at least a 1-grade improvement is evaluated by independent assessor from Baseline using the following scale:
  0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat.
Percentage of Participants Who Achieved a Composite 1-grade Response with Patient-Reported Submental Fat Rating Scale (PR-SMFRS) Compared to the Baseline | Baseline and 12 weeks after last treatment
  The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" answered on a 5-point ordinal scale (0-4):
  0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat.
Change From Baseline in a Magnetic Resonance Imaging (MRI) Response in Pre-platysmal Area | Baseline and 12 weeks after last treatment
  Change rate of reduction in pre-platysmal volume.
Change From Baseline in a Magnetic Resonance Imaging (MRI) Response in Platysmal Area | Baseline and 12 weeks after last treatment
  Change rate of reduction in platysmal volume.
Percentage of Participants Who Achieved a Composite 2-grade Response with Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) Compared to the Baseline | Baseline and 12 weeks after last treatment
  A composite 2-grade response is defined as at least a 2-grade improvement from Baseline on both the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) is evaluated by independent assessor and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) using the following scale:
  0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat.
Change From Baseline in Participants With a Subject Self Rating Scale (SSRS) Response | Baseline and 12 weeks after last treatment
  A SSRS response is defined as an SSRS score that is 4 or greater 12 weeks after the last treatment.
  The SSRS assesses participant's satisfaction with their appearance in association with the face and chin on a 7-point scale from 0 to 6: where 0 = Extremely dissatisfied, 1 = Dissatisfied, 2 = Slightly dissatisfied, 3 = Neither satisfied nor dissatisfied, 4 = Slightly satisfied, 5 = Satisfied and 6 = Extremely satisfied.
Change From Baseline in Patient-Reported Submental Fat Impact Scale (PR-SMFIS) | Baseline and 12 weeks after last treatment
  Patients are asked to rate the visual and emotional impact that the appearance of submental fullness had on their self-perception using 11-point scale range from 0 (no impact) to 10 (extreme impact).
Change From Baseline in Depth of Cervical Mental Angle Analyzed with 3D Scanner | Baseline and 12 weeks after last treatment
  The cervical mental angle is measured using a 3D scanner photograph obtained at first and last visit.
Patient Global Impression of Change scale (PGIC) | 12 weeks after last treatment
  Patient global impression of change scale (PGIC) is to rate patients total improvement or worsening in the appearance since before the first treatment compared to final treatment with 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse.
Change From Baseline in Derriford Appearance Scale 24 (DAS24) | Baseline and 12 weeks after last treatment
  Difference of Derriford Appearance Scale 24 (DAS24) is to measure distress and dysfunction to problems of appearance with 24 questions using 4-point from 0 (None) to 4 (more distress).
Change From Baseline in Body Image Quality of Life Inventory (BIQLI) | Baseline and 12 weeks after last treatment
  Body Image Quality Life Inventory (BIQLI) assesses participants' body image using 7-point ranging from -3 (very negative) to +3 (very positive).

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyeon Lew, MD,PhD, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Yonsei University Health System, Gangnam Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No